CLINICAL TRIAL: NCT03471325
Title: A Comparison of the Outcomes of Two Existing Routine Clinical Therapies for Dental Prophylaxis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National University Health System, Singapore (Other)
Responsible Party: Principal Investigator, Jia Hui Fu, Assistant Professor, National University Health System, Singapore
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2016/00916
Record Dates: First submitted 2018-03-07; First posted 2018-03-20 (Actual); Last update posted 2018-03-21 (Actual); Status verified 2018-03

CONDITIONS: Gingivitis
Keywords: plaque removal
MeSH Terms: conditions — Gingivitis

STUDY DESIGN:
Intervention Model Description: In each subject, his/her right and left dentition will be randomized into Plaque Disclosed (PD) and Non Plaque Disclosed (NPD) groups. Subsequently, the upper and lower jaws will be randomized into Air Flow (AF) and Rubber Cup (RC).
Who Masked: Participant, Outcomes Assessor
Masking Description: The examiner, who chart the plaque score is blinded to the treatment assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Plaque Disclosed with Air Flow (PDAF) (Experimental): Plaque will be disclosed prior to polishing with the air flow system.
  Interventions: Procedure: Plaque disclosed with air flow
- Plaque Disclosed with Rubber Cup (PD-RC) (Experimental): Plaque will be disclosed prior to polishing with the rubber cup and fine grit prophylaxis paste.
  Interventions: Procedure: Plaque disclosed with rubber cup
- Non Plaque Disclosed Air Flow (NPD-AF) (Experimental): Air polishing system will be used to remove the plaque
  Interventions: Procedure: Non plaque disclosed air flow
- Non Plaque Disclosed Rubber Cup (NPD-RC) (Placebo Comparator): Rubber Cup polishing to remove plaque.
  Interventions: Procedure: Non plaque disclosed rubber cup

INTERVENTIONS:
Procedure: Plaque disclosed with air flow — air polishing with prior plaque disclosing
  Other Names: EMS
  Arms: Plaque Disclosed with Air Flow (PDAF)
Procedure: Plaque disclosed with rubber cup — rubber cup polishing with prior plaque disclosing
  Other Names: Slow speed handpiece
  Arms: Plaque Disclosed with Rubber Cup (PD-RC)
Procedure: Non plaque disclosed air flow — air polishing with no prior plaque disclosing
  Other Names: EMS
  Arms: Non Plaque Disclosed Air Flow (NPD-AF)
Procedure: Non plaque disclosed rubber cup — rubber cup polishing with no prior plaque disclosing
  Other Names: Slow speed handpiece
  Arms: Non Plaque Disclosed Rubber Cup (NPD-RC)

SUMMARY:
Background: In most practices, conventional in-office prophylaxis starts immediately with scaling and polishing. Therefore, this project was designed to challenge tradition by comparing plaque removal efficacy of rubber cup and air polishing in two scenarios, one where plaque was disclosed prior to treatment and the other where plaque was not disclosed.

Methods: In this randomized, single blind, split-mouth design clinical trial, healthy, non-smoking participants with poor oral hygiene were recruited. Quadrants in each participant were randomly assigned to 4 treatment groups, which were plaque disclosure with rubber cup polishing, no plaque disclosure with rubber cup polishing, plaque disclosure with air polishing, and no plaque disclosure with air polishing. Examiners were calibrated and masked to the treatment rendered in each quadrant. Post treatment satisfaction questionnaires for both participants and operators were completed. Plaque scores for each quadrant and treatment time were the recorded outcome measures.

DETAILED DESCRIPTION:
According to the literature search, there was no preceding study, which compared the efficacy of conventional routine of rubber cup or air powder polishing with or without prior plaque disclosure. Therefore, this study was designed to test the hypotheses that (1) disclosing plaque prior to dental polishing was more effective than dental polishing alone, (2) air polishing was more efficient than rubber cup polishing, and (3) operators and patients prefer air polishing to rubber cup polishing.

In order to evaluate the hypotheses raised, a single blind, randomised controlled clinical trial with a split mouth design was conducted. The control groups had conventional dental prophylaxis regime of mechanical plaque removal with either fine air powder polishing or rubber cup polishing using fine grit prophylaxis paste. The test groups had plaque disclosure prior to mechanical plaque removal as described for the control groups. In total, there were 4 study groups: (1) rubber cup polishing without prior plaque disclosure (RC-NPD) (negative control), (2) rubber cup polishing with prior plaque disclosure (RC-PD) (positive control), (3) air polishing without prior plaque disclosure (AF-NPD) (negative test), and (4) air polishing with prior plaque disclosure (AF-PD) (positive test).

The quadrant that was assigned to receive RC-NPD was treated first followed by the quadrant assigned to receive AF-NPD. Plaque was disclosed in all 4 quadrants and the assigned calibrated examiner proceeded to chart the FMPS. Next, the quadrant assigned to receive RC-PD was treated, followed by the quadrant assigned to receive AF-PD; subsequently FMPS was charted. Any aberrant findings in occlusion, tooth alignment, extra/missing teeth were also noted. A digital stopwatch was used to time the treatment duration for each quadrant. Both participant and clinician completed a post prophylaxis satisfaction questionnaire. The treatment workflow used in this study was illustrated in figure 1. The primary outcome measure was the post treatment FMPS and the secondary outcomes measures were the treatment duration.

Descriptive statistics (mean and standard deviations) was used to summarize the plaque score and treatment duration for each study group. Two-way repeated measure ANOVA test was employed to examine the study hypotheses that air polishing was more effective in removing plaque compared to rubber cup polishing and disclosing plaque prior to prophylaxis increased the thoroughness of the prophylaxis. Two-way repeated measure ANOVA test was also performed to study the treatment duration between the 2 polishing methods and treatment regimens of with or without plaque disclosure prior to prophylaxis. In a secondary analysis, interactions were tested to study if there were differences among the 4 operators. Paired T-test and Pearson's Chi-Square tests were used to study the participant's and operator's preference for each treatment modality based on various yardsticks and overall, respectively. The level of significance was set at p-value<0.05. All statistical analyses were carried out using a statistical package.

ELIGIBILITY:
Inclusion Criteria:

* 1) Age 21 to 35 years old
* 2) Healthy
* 3) Non-smoker
* 4) With gingivitis and poor oral hygiene (plaque score of at least 50%)
* 5) English literate

Exclusion Criteria:

* 1) Smoker
* 2) Pregnant or lactating females
* 3) Unable to speak/read/write/communicate in English
* 4) With dentures or bridges or braces

Ages: 21 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 89 (Actual)
Dates: Start 2016-12-08 (Actual); Primary Completion 2017-09-30 (Actual); Study Completion 2017-12-14 (Actual)

PRIMARY OUTCOMES:
post treatment plaque score | 1 day
  plaque score based on Loe and Silness 1963. Minimum score is 0. Maximum score is 1. It is a categorical scale of 0 or 1 and is not a continuous scale.
  0 is a good outcome and 1 is a poor outcome. Each side of the tooth will be recorded as either a 0 or a 1. It will be added up and averaged out by the number of tooth sides multiple by 100% to get a percentage total score. The higher the percentage, the worser the outcome.

SECONDARY OUTCOMES:
Treatment duration | 1 day
  Time taken to complete the polishing by the air flow system or rubber cup polishing

CONTACTS AND LOCATIONS:
Overall Officials: Jia Hui Fu, Principal Investigator — National University Health System, Singapore

IPD SHARING:
Plan to Share IPD: No